CLINICAL TRIAL: NCT01015274
Title: Non-invasive Assessment of Skeletal Muscle Loss in Cancer Patients
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 09-150; 1R43AR054993-01A,; AR054993; 1R43AR054993-01 (NIH)
Record Dates: First submitted 2009-11-16; First posted 2009-11-18 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2011-07

CONDITIONS: Cachexia
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy control male

SUMMARY:
The long-term objective of this research is to develop a non-invasive approach for early assessment of which patients are at high risk for future development of skeletal muscle atrophy. The investigators hypothesize that the rate constant for the terminal portion of the isotope decay curve following ingestion of a single oral dose of deuterated-3-methylhistidine (D-3MH) provides an accurate measure of this increased risk and that this rate constant can be measured non-invasively from timed spot urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 30-75 years old
* Body Mass Index (BMI) <27 kg/m2

Exclusion Criteria:

* Uncontrolled hypertension
* Glomerular filtration rate less than 60 mL/min/1.73 m2
* History of recurrent gastrointestinal bleeding
* Unable or unwilling to provide informed consent
* Ongoing anti-coagulant therapy

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample of healthy males
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2009-10

CONTACTS AND LOCATIONS:
Overall Officials: Morteza Janghorbani, Ph.D., Principal Investigator — BIOCHEMANALYSIS CORPORATION; Melinda Sheffield-Moore, Ph.D., Study Director — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States